CLINICAL TRIAL: NCT01317459
Title: Using Guided Self-determination (GSD) to Promote Improved Self-management in Adults With Type 1 Diabetes - an Intervention Study.
Brief Title: Guided Self-determination - Promoting Self-management in Type 1 Diabetes
Acronym: GSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010/1325
Record Dates: First submitted 2011-03-11; First posted 2011-03-17 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes
Keywords: Self management; Diabetes type one; Empowerment; Intrinsic motivation
MeSH Terms: conditions — Diabetes Mellitus; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counselling (Experimental)
  Interventions: Behavioral: Guided self-determination
- No intervention (Experimental): Care as usual
  Interventions: Behavioral: Guided self-determination

INTERVENTIONS:
Behavioral: Guided self-determination — Group counselling

SUMMARY:
Background: 50% of people with diabetes are living with too high blood sugars and increased risk of diabetes related complications together with poor quality of life. The need to improve diabetes care by better enabling patients to utilise their individual and local resources to self-manage the condition is widely recognized, yet there is a lack of access to evidence-based patient-centred healthcare interventions. At present the individual patient's judgement of own concrete situation mostly remains unexplored and insufficiently used in decision-making causing that problems perceived by the patient in living with the illness remain unrecognised and insufficiently resolved.

Aim and Methods: Guided self-determination (GSD) is an educational method developed to promote patient autonomy, participation, skills building and intrinsic motivation. In this evidence-based group-intervention the main objective is to implement and evaluate GSD through a randomised controlled trial. GSD methods will be performed seven times for the intervention group. The control group will receive traditional out-patient consultations - 'care as usual' Outcome measures will be performed at baseline, after 9 and 18 months. The project will focus on adults with type 1 diabetes (18-55 yrs) where an improvement will be highly cost-effective in preventing late complications and enhanced psychosocial health. GSD is presumably an intervention providing psychosocial support applicable in busy clinical practice.

An alliance is established between Haukeland University Hospital, Norway and Steno Diabetes centre, Copenhagen, Denmark, Centre of Evidence-Based Practice, Bergen University College, and Bergen University to conduct this intervention and thus make the best possible use of interrelated knowledge within the issue.

ELIGIBILITY:
Inclusion Criteria:

Diabetes type one, HbA1c >= 8%

Exclusion Criteria:

Pregnancy, decreased cognitive function and/or serious mental health disturbances, language barriers to the Norwegian language

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 0, 9 and 18 months

SECONDARY OUTCOMES:
Who 5 | 0, 9 and 18 months
TSRQ scales | 0, 9 and 18 months
PAID scales | 0, 9 and 18 months
Rosenberg's self-esteem scale | 0, 9 and 18 months
PCD scales | 0, 9 and 18 months
HCCQ scales | 0, 9 and 18 months
DDS scales | 0, 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marit Graue, RN, PhD, Principal Investigator — Bergen University College
Locations (1):
- Helse Vest HF, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Mohn J, Igland J, Zoffmann V, Peyrot M, Graue M. Factors explaining variation in self-esteem among persons with type 1 diabetes and elevated HbA1c. PLoS One. 2018 Aug 10;13(8):e0201006. doi: 10.1371/journal.pone.0201006. eCollection 2018. PMID 30096144
- [Derived] Mohn J, Graue M, Assmus J, Zoffmann V, Thordarson H, Peyrot M, Rokne B. The effect of guided self-determination on self-management in persons with type 1 diabetes mellitus and HbA1c >/=64 mmol/mol: a group-based randomised controlled trial. BMJ Open. 2017 Jul 3;7(6):e013295. doi: 10.1136/bmjopen-2016-013295. PMID 28674125